CLINICAL TRIAL: NCT05473650
Title: A Spectrum of Hematological Disorders in Children Presented With Pancytopenia at Assiut University Hospital
Brief Title: Spectrum of Hematological Disorders in Pediatrics
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Zakria Younes Mohammed Essemy, resident doctor, Assiut University
Other Study IDs: pancytopenia in pediatrics
Record Dates: First submitted 2022-07-19; First posted 2022-07-26 (Actual); Last update posted 2022-07-26 (Actual); Status verified 2022-07

CONDITIONS: Pancytopenia
MeSH Terms: conditions — Pancytopenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: CBC.with with differential Peripheral smear — determine spectrum of hematological disorders in childern with pancytopenia

SUMMARY:
To determine the spectrum of pancytopenia with its frequency and etiology in children presenting to Assiut University Children Hospital during one year

DETAILED DESCRIPTION:
Pancytopenia is a condition in which there is a decrease of all the three cellular elements of blood, namely erythrocytes, leukocytes, and platelets . It is quite a common finding among children. According to regional studies, it makes up around 2.90% to 3.57% of the burden of presentations in the pediatric population. Some of the presenting symptoms include, but are not limited to, pallor, fever, weight loss, dyspnea, bleeding, bruising, visceromegaly, and increased risk of infections .

Pancytopenia is not a disease in itself but a laboratory finding of the constitution of diseases. It can occur due to a variety of disorders which can be as simple as nutritional deficiencies to serious malignant disorders . Megaloblastic anemia and acute lymphoblastic leukemia are among the most common presentations of pancytopenia.

Pancytopenia results in a hypoplastic bone marrow. It is diagnosed on the basis of the complete blood count test. Pancytopenia is labeled when the hemoglobin (hb) is less than 10 gm%, absolute neutrophil count (anc) is less than 1.5*109/l, and platelet count is less than 100*109/l [9].

But, in order to find out the etiological factor causing pancytopenia, bone marrowexamination is done. Being an interventional procedure, it is relatively safe with little or no risk of bleeding.

Etiology of pancytopenia The etiology of pancytopenia can be broadly categorized as a central type that involves disorders of production or a peripheral type that involves disorders of increased destruction.These causes could contribute to the pancytopenia independently or as a combination.

Decreased production (central type): Pancytopenia due to decreased production is mostly secondary to nutritional deficiencies. Pancytopenia caused by bone marrow failure is known as aplastic anemia. Aplastic anemia could be idiopathic/autoimmune, secondary to infections (such as parvovirus B19, hepatitis, human immunodeficiency virus (HIV), cytomegalovirus, or Epstein-Barr virus), after drug toxicity, or chemotherapeutic agents (methotrexate, dapsone, carbimazole, carbamazepine, chloramphenicol). Pancytopenia can also be related to inadequate intake (as seen in eating disorders and alcoholics) or malabsorption.The production of cell lines is also impaired when the bone marrow is infiltrated by malignancies (lymphoma, leukemia, multiple myeloma) or granulomatous disorders. Metastatic tumors can also cause bone marrow replacement late in the disease, thus producing pancytopenia.

Increased destruction (peripheral type): Peripheral destruction of cells can be associated with many autoimmune conditions (such as systemic lupus erythematosus, rheumatoid arthritis) and splenic sequestration (alcoholic liver cirrhosis, HIV, tuberculosis, malaria). Hypersplenism affects more frequently the platelets and erythrocytes than leukocytes.

Differential diagnosis Multiple conditions can present with pancytopenia; hence, when someone shows with pancytopenia, a complete evaluation is performed to detect the cause of pancytopenia. Bone marrow disorders such as aplastic anemia, myelodysplastic syndrome, acute leukemia, myelofibrosis, megaloblastic anemia, paroxysmal nocturnal hemoglobinuria, and Fanconi's anemia can present with pancytopenia. Fanconi anemia is the most common congenital cause of bone marrow failure with an autosomal recessive inheritance pattern. In myelofibrosis, there is a replacement of the bone marrow cells with fibrotic tissue. Malignancies such as lymphoma, multiple myeloma, and hairy cell leukemia can also present with pancytopenia. Non-bone marrow conditions present with pancytopenia include systemic lupus erythematosus, infections (such as parvovirus B19, Epstein Barr virus, HIV, hepatitis, leishmaniasis, tuberculosis, malaria, and histoplasmosis).

ELIGIBILITY:
Inclusion Criteria:

* All patients with presistant pancytopenia from age 1 month to 18 years at Assiut university hospital of pediatrics

Exclusion Criteria:

* Patients below age of 1 month or above 18 years

Ages: 28 Days to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: patients with pancytopenia from the age of one month to 18 years old
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-09-01 (Estimated); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-11-01 (Estimated)

PRIMARY OUTCOMES:
percentage of aplastic anemia among other causes of pancytopenia in childern presented to assiut university childern hospital with abnormal CBC | one year
  getting a proper diagnosis of different cases of pancytopeina in childern which helps in their treatment

REFERENCES:
- [Background] Memon S, Shaikh S, Nizamani MA. Etiological spectrum of pancytopenia based on bone marrow examination in children. J Coll Physicians Surg Pak. 2008 Mar;18(3):163-7. PMID 18460245
- [Background] Sharma R, Nalepa G. Evaluation and Management of Chronic Pancytopenia. Pediatr Rev. 2016 Mar;37(3):101-111; quiz 112-3. doi: 10.1542/pir.2014-0087. No abstract available. PMID 26933225
- [Background] Das Makheja K, Kumar Maheshwari B, Arain S, Kumar S, Kumari S, Vikash. The common causes leading to pancytopenia in patients presenting to tertiary care hospital. Pak J Med Sci. 2013 Sep;29(5):1108-11. doi: 10.12669/pjms.295.3458. PMID 24353701
- [Background] Zeb Jan A, Zahid B, Ahmad S, Gul Z. Pancytopenia in children: A 6-year spectrum of patients admitted to Pediatric Department of Rehman Medical Institute, Peshawar. Pak J Med Sci. 2013 Sep;29(5):1153-7. doi: 10.12669/pjms.295.3865. PMID 24353710
- [Background] Jain A, Naniwadekar M. An etiological reappraisal of pancytopenia - largest series reported to date from a single tertiary care teaching hospital. BMC Hematol. 2013 Nov 6;13(1):10. doi: 10.1186/2052-1839-13-10. PMID 24238033
- [Background] Gnanaraj J, Parnes A, Francis CW, Go RS, Takemoto CM, Hashmi SK. Approach to pancytopenia: Diagnostic algorithm for clinical hematologists. Blood Rev. 2018 Sep;32(5):361-367. doi: 10.1016/j.blre.2018.03.001. Epub 2018 Mar 5. PMID 29555368
- [Background] Takeshima M, Ishikawa H, Kitadate A, Sasaki R, Kobayashi T, Nanjyo H, Kanbayashi T, Shimizu T. Anorexia nervosa-associated pancytopenia mimicking idiopathic aplastic anemia: a case report. BMC Psychiatry. 2018 May 25;18(1):150. doi: 10.1186/s12888-018-1743-6. PMID 29801443